CLINICAL TRIAL: NCT02029339
Title: Continuous Topical Triple-tube Instillation and Suction for for Open Abdomen in the Septic Patients With Complicated Intra-abdominal Infections
Brief Title: Continuous Topical Instillation for Open Abdomen in the Septic Patients With Complicated Intra-abdominal Infections
Acronym: Triple-tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Qingsong Tao, Attending Surgeon, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81000153
Record Dates: First submitted 2013-12-28; First posted 2014-01-07 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-01

CONDITIONS: Wound Infection
Keywords: Negative pressure wound therapy; Acute wound infection; complicated abdominal infection; Cytokines; Matrix metalloproteinase
MeSH Terms: conditions — Wound Infection | interventions — Suction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triple-tube group (Experimental): The patients were treated with continuous topical triple-tube irrigation and suction
  Interventions: Device: Continuous topical triple-tube irrigation and suction
- SOC group (Active Comparator): The patients were treated with standard of care (SOC) without topical irrigation
  Interventions: Device: SOC

INTERVENTIONS:
Device: Continuous topical triple-tube irrigation and suction — The triple-tube device was continuous operated: instilled the topical solution through the "washing tube", delivered negative pressure therapy at 100 - 125 mmHg continuously through the inner tube of "sleeve tubes" through the central negative pressure device in the wall of the ward. The outer tube was used for normalize and balance the distribution of the negative pressure around the inner tube to allow the solution to penetrate through the dressing to cover the wound, and protecting the inner tube from getting stuck with the sucked tissue. All tubes are all commercially available (Medical Silicone Tubing, Forbest Manufacturing Co., Ltd, China).
  Arms: triple-tube group
Device: SOC — Debridement, offloading, standard moist wound care, and conventional NPWT without continuous irrigation are the fundamental SOC for Open Abdomen with complicated abdominal infections.
  Other Names: standard of care
  Arms: SOC group

SUMMARY:
The closed systems, such as conventional negative pressure wound therapy (NPWT), were usually avoided in infected or critical colonized wounds. To our observation, the additional continuous irrigation tube attached beside the suction tube in the NPWT system could provide the effective drainage by reducing the occlusion of suction tube, enable effective debridement by diluting infected/necrotized tissues and decrease the incidence of fistula by providing relatively moist ambient. At our institutions, the modified system combined with a "triple-tube" device to allow a continuous instillation became more active and efficient. The study is to investigate if a continuous triple-tube instillation and suction could improve the outcomes of acute severely infected open abdomen.

DETAILED DESCRIPTION:
This study was performed on the patients with a severely complicated infected open abdomen treated with topical triple-tube irrigation and suction, compared with a control group of the patients treated with standard NPWT without topical irrigation. The clinical outcomes were recorded. Profiles of cytokines/proteinase in wound fluid were quantified weekly.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years patients with complicated intra-abdominal infections who needed open abdomen (OA) and vacuum-assisted wound closure and mesh-mediated fascial traction (VAWCM)
* Eligible patients were properly consented before enrollment. If the patient was incapable, the patient's legal representative was asked to provide consent on the patient's behalf.
* Patients with grade 1b (contaminated OA without adherence between bowel and abdominal wall), 2b (contaminated OA developing adherence) open abdomen, as classified by Bjorck.

Exclusion Criteria:

* < 18 years,
* pre-existing large ventral hernia
* Frozen OA with adherent bowel (OA of grade 4),
* Clean wound (OA of grade 1a or 2a)
* chronic wound infection
* critical wound ischemia
* severe systemic infection
* end-stage renal disease
* severe liver disease
* uncontrolled diabetes mellitus
* any issue with an obviously high risk of delayed wound healing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Delayed primary fascial closure | Up to 8 weeks
  Delayed primary fascial closure, Time to infection clearance and abdomen closure, ICU and hospital length of stay

SECONDARY OUTCOMES:
Levels of cytokines/proteinase in wound fluid | Up to 8 weeks
  Wound fluid was collected at the initial admission and every three days later. Before samples were collected, irrigation was released and held for 6 hours to avoid contamination or dilution by the washed solution. Wound fluid was collected using a filter paper (PerioPaper, Oraflow Inc., NY) for 30 seconds as prior described and stored at -80°C until analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Qingsong Tao, MD, PhD, Principal Investigator — Department of Surgery, Zhongda Hospital, Southeast University Medical School
Locations (1):
- Department of Surgery, Zhongda Hospital, Southeast University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Gabriel A, Shores J, Heinrich C, Baqai W, Kalina S, Sogioka N, Gupta S. Negative pressure wound therapy with instillation: a pilot study describing a new method for treating infected wounds. Int Wound J. 2008 Jun;5(3):399-413. doi: 10.1111/j.1742-481X.2007.00423.x. PMID 18593390
- [Background] Vuerstaek JD, Vainas T, Wuite J, Nelemans P, Neumann MH, Veraart JC. State-of-the-art treatment of chronic leg ulcers: A randomized controlled trial comparing vacuum-assisted closure (V.A.C.) with modern wound dressings. J Vasc Surg. 2006 Nov;44(5):1029-37; discussion 1038. doi: 10.1016/j.jvs.2006.07.030. Epub 2006 Sep 26. PMID 17000077
- [Background] Fluieraru S, Bekara F, Naud M, Herlin C, Faure C, Trial C, Teot L. Sterile-water negative pressure instillation therapy for complex wounds and NPWT failures. J Wound Care. 2013 Jun;22(6):293-4, 296, 298-9. doi: 10.12968/jowc.2013.22.6.293. PMID 24049811
- [Background] Lessing MC, James RB, Ingram SC. Comparison of the Effects of Different Negative Pressure Wound Therapy Modes-Continuous, Noncontinuous, and With Instillation-on Porcine Excisional Wounds. Eplasty. 2013 Oct 1;13:e51. eCollection 2013. PMID 24106564